CLINICAL TRIAL: NCT01801852
Title: Phase 1 Study of Autologous Natural Killer T Cells Infusion in Treating Patients With Tumors
Brief Title: Autologous Natural Killer T Cells Infusion for the Treatment of Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Tsinghua University (Other)
Responsible Party: Principal Investigator, Han weidong, PI, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-003
Record Dates: First submitted 2013-02-22; First posted 2013-03-01 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer; Glioma; Hepatocellular Cancer; Squamous Cell Lung Cancer; Pancreatic Cancer; Colon Cancer; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Glioma; Liver Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NKT cells (Experimental): NKT cells treatment plus regular treatment
  Interventions: Biological: NKT cells

INTERVENTIONS:
Biological: NKT cells

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of natural killer T (NKT) cell-based autologous adoptive immunotherapy in subjects with metastatic, treatment-refractory breast cancer, glioma, hepatocellular carcinoma, squamous cell lung cancer, pancreatic cancer, colon cancer or prostate cancer.

DETAILED DESCRIPTION:
A randomized controlled trial on the efficacy and safety of autologous natural killer T (NKT) cells infusion treatment in advanced cancer.

ELIGIBILITY:
Inclusion Criteria:•Male or female not less than 18 years of age or over 80 years of age.

* Life expectancy of ≥ 24 weeks as measured by the Eastern Cooperative Oncology Group (ECOG) performance status.
* Subjects must present with one of the following disease pathologies: Breast Cancer, Glioma, Hepatocellular Cancer, Squamous Cell Lung Cancer, Pancreatic Cancer, Colon Cancer or Prostate Cancer
* The pathology must be an assessable disease (measurable by CT scan or MRI) that is refractory to standard treatments (e.g., chemotherapy, radiation, etc.)
* Negative for hepatitis B, hepatitis C, HIV, and CMV.
* Subjects must present with leukocyte counts above 3,000/μL and platelet counts above 100,000/ μL.
* Subjects must present with minimum hemoglobin levels of 10.
* If female, subject is surgically sterile (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), post menopausal (no menses >12 months), or using a high-efficiency method of contraception such as implant, injectable, combination oral contraceptive, intrauterine device (IUD) or sexual abstinence, or has a vasectomized partner.
* If female of childbearing potential, subject is not pregnant, breast-feeding or planning a pregnancy during the study, and has a negative pregnancy test on screening visit.
* Able to comprehend and sign an informed consent document and comply with the requirements of the study.

Exclusion Criteria:•No measurable malignant disease by CT scan or tumor markers.

* Life expectancy of ≤ 24 weeks as measured by the Eastern Cooperative Oncology Group (ECOG) performance status.
* Age of less than 18 years or over 80 years of age.
* Documented/confirmed positive testing for hepatitis B, hepatitis C, HIV, or CMV.
* Prior or current history of autoimmune disease.
* Pregnant or lactating women.
* Leukocyte count < 3,000 /μL prior to leukapheresis.
* Platelet count < 100,000/μL prior to leukapheresis.
* Hemoglobin levels below 10.
* PTT (prothrombin time) of < 12 seconds or > than 15 seconds.
* aPTT (activated partial thromboplastin time) of < 25 seconds or > than 39 seconds.
* Failure or refusal to sign informed consent for the study.
* Culture fails to meet specifications for study.
* Subject has any other medical condition that, in the opinion of the investigator, might significantly affect the ability to safely participate in the study or affect the conduct of the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-05 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | Until week 24
  defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment

SECONDARY OUTCOMES:
Anti-tumor responses to NKT cells infusions | at least once within 30 days afther completing four-cycle treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China